CLINICAL TRIAL: NCT01400035
Title: The Investigation of Vinpocetine (Cavinton) for Treatment of Acute Cerebral Infarction, an Open, Multicenter, Randomized, Control Study
Brief Title: Chinese Assessment for Vinpocetine In Neurology
Acronym: CAVIN
Status: Completed | Type: Observational
Sponsor: Shanghai Rxmidas Pharmaceuticals Co. Ltd. (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Principal Investigator, Weiwei Zhang, Director of Neurology Department, Shanghai Rxmidas Pharmaceuticals Co. Ltd.
Other Study IDs: RMS2010C
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Cerebral Infarction
Keywords: acute cerebral infarction, Vinpocetine
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- test group, control group: Test group: Patients will be given cytidine diphosphate choline 0.4-0.5g, aspirin 75-100mg or Clopidogrel 75mg, intravenous infusion of Cavinton 30mg once a day.
  Control group: Patients will be given cytidine diphosphate choline 0.4-0.5g, aspirin 75-100mg or Clopidogrel 75mg once a day.

SUMMARY:
Trial Title：The treatment of Vinpocetine（Cavinton）in patients with cerebral infarction, an open, randomized, multi-center control study

1. Objectives Evaluate the efficacy and safety of Vinpocetine（Cavinton）for treatment of cerebral infarction
2. Design Open, randomized, multi-center control study
3. Trial Population:Patients with acute cerebral infarction
4. Number of Subjects 720 patients in test group and 240 patients in control group, totally 960 patients will be recruited.
5. Administration Test group: intravenous infusion drip of Vinpocetine 30 mg and Citicoline 0.4g once daily; additionally oral take aspirin 75-100mg or clopidogrel sulfate tablets 75mg once a day.

   Control group: intravenous infusion drip of Citicoline 0.4g once daily; additionally oral take aspirin 75-100mg or clopidogrel sulfate tablets 75mg once a day.
6. Outcome evaluation 6.1 Primary end points: 6.1.1 Modified Rankin Scale. 6.1.2 Mini-Mental State Examination (MMSE) 6.2 Second end points 6.2.1 Barthel index 6.2.2 NIHSS score 6.2.3 Transcranial Doppler (TCD) examination 6.3 Safety data 6.3.1 Serology, hepatic and renal function examination 6.3.2 Adverse events
7. Statistical Analysis: SPSS 11.0 will be used to make the data analysis.

DETAILED DESCRIPTION:
The design of this study is a randomized, open, multi-center and control study. The patients with cerebral infarction are as the study objects. Coronal CT / MRI examination combined with NIHSS and Modified Ranking Scale, MMSE, Barthel index, Transcranial Doppler (TCD) examination are applied to evaluate the Vinpocetine treatment efficacy and safety for cerebral infarction [14]. From ethical side, all patients will receive a conventional therapy, and based on it, the test group will be given intravenous injection of Vinpocetine as add-on treatment. Observation period is 10-14 days, and follow up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 40-80
* The onset of the infarction between 48 hours and 1 month
* CT / MRI results show cerebral infarction with deficit of neurological function.
* CT or MRI confirms no intracranial hemorrhage
* NIHSS score ≥ 3
* The subject agree to sign the informed consent form

Exclusion Criteria:

* Evidence of acute or chronic intracranial hemorrhage, subarachnoid hemorrhage, intracranial arteriovenous malformation, aneurysm or neoplasm based on CT / MRI examination
* NIHSS score ≥ 17
* Coma patient
* Existed disorders or conditions that would interfere neurological assessments (eg. dementia, psychiatric disorder, etc.)
* Intracranial tumor, arteriovenous malformation, aneurysm, or intracranial surgery
* Active peptic ulcer disease
* Complicated with severe hepatic and renal disorder (ALT, AST 3.0 times higher than normal value; BUN or Cr more than 1.5 times the normal value) and severe disorder in hematopoietic system and endocrine system.
* Bleeding tendency or blood disease
* Plan to perform operation and carotid angioplasty
* With severe congestive heart failure or acute myocardial infarction
* Participate in other clinical trials at the same time, or withdrawal within 3 months
* Allergic or contraindicated to vinpocetine or other treatment medication
* Investigator think the subject is not suitable to participate in this trial

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Totally 610 subjects were recruited, 469 in test group and 141 in control group.
Sampling Method: Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE)and Modified Rankin Scale | May 2010 - Feb. 2013

SECONDARY OUTCOMES:
Barthel index and NIHSS | May. 2010 - Feb. 2013

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Zhang, MD, Principal Investigator — PLA.The Military General Hospital of Beijing
Locations (1):
- Weiwei Zhang, Beijing, China